CLINICAL TRIAL: NCT00286780
Title: A Phase 2, Open Label Study of AT-101 in Combination With Rituximab in Patients With Relapse or Refractory Chronic Lymphocytic Leukemia
Brief Title: Phase 2 Safety and Efficacy Study of AT-101 in Combination With Rituximab in Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascenta Therapeutics (Industry)
Responsible Party: Brian Wood, Associate Director, Clinical Development, Ascenta Therapeutics
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AT-101-CS-008
Record Dates: First submitted 2006-02-03; First posted 2006-02-06 (Estimated); Last update posted 2010-08-13 (Estimated); Status verified 2010-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: AT101; AT-101; cancer; lymphoctic; lukemia; Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms | interventions — gossypol acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: AT-101

INTERVENTIONS:
Drug: AT-101 — 80 mg of AT-101 once daily for three days every other week, 375 mg/m2 of rituximab weekly for up to 12 weeks

SUMMARY:
This is an open-label Phase 2 study to evaluate the safety and efficay of AT-101 in combination with rituximab in patients with relapsed or refractory chronic lymphocytic leukemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL as defined by the NCI-working group
* Previous treatment with standard systemic chemotherapy or immunotherapy.
* Disease progression or relapse after treatment.
* Indication for treatment as defined by the NCI Working Group Guidelines (Cheson, 1996)
* ECOG performance status ≤ 2
* Adequate liver and renal and bone marrow function

Exclusion Criteria:

* Treatment of CLL with chemotherapy, monoclonal antibody or radiotherapy within 60 days prior to entering the study. Acute toxicities from prior therapy must have resolved to Grade ≤ 1.
* Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Severe or debilitating pulmonary disease (dyspnea at rest, significant shortness of breath, COPD)
* Active secondary malignancy or history of other malignancy within the last five years
* Active symptomatic fungal, bacterial and/or viral infection including active HIV or viral hepatitis (A, B or C).
* Patients who are contraindicated for treatment with rituximab
* Diagnosis of prolymphocytic leukemia, hairy cell leukemia, leukemic phase of non-Hodgkin's lymphoma, or other non-B-CLL B-cell malignancy;
* T-CLL or other T-cell malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2006-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Safety of AT-101 in combination with rituximab | 5 months for each patient; 20 months entire study

SECONDARY OUTCOMES:
Preliminary efficacy of AT-101 in combination with rituximab | 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kipps, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, San Diego, California, United States